CLINICAL TRIAL: NCT07317752
Title: Incidenza Della Disgeusia Nei Pazienti Affetti da Carcinoma Mammario in Trattamento Chemioterapico: Uno Studio Pilota Prospettico
Brief Title: Incidence of Dysgeusia in Breast Cancer Patients Undergoing Chemotherapy
Acronym: GustiAmo
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Sanitaria Locale CN2 Alba-Bra (Other)
Responsible Party: Sponsor
Other Study IDs: GustiAmo
Record Dates: First submitted 2025-12-05; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Taste Disorders; Breast Cancer; Quality of Life; Taste Perception; Dysgeusia; Chemotherapy Effects; Nutritional Status; Sensory Testing
Keywords: Dysgeusia; Taste disorders; Breast cancer; Quality of life; Taste perception; Chemotherapy effects; Nutritional status; Sensory testing
MeSH Terms: conditions — Taste Disorders; Breast Neoplasms; Dysgeusia | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-Metastatic Breast Cancer Patients Receiving Chemotherapy: This group includes male and female participants diagnosed with non-metastatic breast cancer who are receiving neoadjuvant or adjuvant chemotherapy according to standard clinical practice. All participants are treated at the Oncology Unit of Michele and Pietro Ferrero Hospital in Verduno. Eligible participants are those for whom chemotherapy is indicated as part of routine care and who are willing and able to complete sensory tests, nutritional assessments, and quality-of-life questionnaires during the study period.
  Interventions: Other: Taste Assessment / Nutritional Assessment / Quality of Life Assessment

INTERVENTIONS:
Other: Taste Assessment / Nutritional Assessment / Quality of Life Assessment — Participants will undergo additional procedures as part of the study to assess taste function, nutritional status, and quality of life. These procedures include:
  * Taste assessment using standardized taste strips to measure recognition thresholds for the five basic tastes (sweet, sour, salty, bitter, umami) and chemesthetic sensitivity using strips impregnated with capsaicin.
  * Questionnaires to evaluate chemotherapy-induced taste alterations (CiTAS) and general quality of life (FACT-G).
  * Nutritional assessment, including evaluation of caloric and macronutrient intake using 24-hour dietary recalls, assessment of nutritional status according to GLIM criteria, and measurement of phase angle through bioelectrical impedance analysis (BIA).
  All procedures are non-invasive and performed in addition to the participants' standard chemotherapy treatment.

SUMMARY:
The goal of this observational study is to examine how frequently changes in taste occur in people with early-stage breast cancer who receive chemotherapy. It will also look at how these taste changes affect nutrition and quality of life. The main questions this study aims to answer are:

* How many participants develop changes in taste during chemotherapy?
* How do these changes affect eating habits, nutrition, and daily life?

Participants are women with non-metastatic breast cancer who are receiving chemotherapy before or after surgery.

Researchers will use standardized taste tests to measure how well participants can perceive different flavors. These tests are designed to provide accurate and reproducible results.

Participants will:

* Take part in taste tests during their chemotherapy treatment
* Have their nutritional status evaluated
* Answer questions about their quality of life

DETAILED DESCRIPTION:
Dysgeusia, defined as an altered perception of taste, is a frequent but understudied adverse effect of several chemotherapy regimens used for the treatment of breast cancer. Taste alterations may arise from direct cytotoxic effects on taste receptor cells, changes in saliva composition, mucosal inflammation, altered signal transduction, or central nervous system effects. These disturbances can lead to reduced food enjoyment, alterations in dietary patterns, and potential deterioration of nutritional and functional status.

Although dysgeusia is commonly reported in clinical practice, estimates of its prevalence vary widely due to heterogeneous methodologies and the predominant reliance on self-reported symptoms rather than standardized sensory testing. Studies that objectively quantify changes in taste recognition thresholds during chemotherapy are limited, and little is known about specific aspects such as umami perception or chemesthetic sensitivity. Furthermore, factors that may predispose individual patients to developing dysgeusia-such as baseline taster status, nutritional condition, or specific treatment characteristics-remain poorly characterized.

This observational pilot study was designed to provide objective, reproducible data on taste function in patients with non-metastatic breast cancer receiving standard neoadjuvant or adjuvant chemotherapy. A combination of validated sensory tools, including taste strips and chemesthetic tests, is used to measure changes in taste perception over the course of treatment. Standardized methods were selected to ensure high sensitivity and repeatability and to allow quantitative comparison across different time points.

The study also integrates nutritional assessment and quality-of-life evaluation to explore the broader clinical implications of dysgeusia. Particular attention is given to potential associations between objective taste alterations, patient-reported symptoms, and parameters such as nutritional status, dietary intake, and functional well-being. Given the scarcity of comprehensive, methodologically rigorous studies in this area, the data generated may help clarify the clinical burden of dysgeusia and inform strategies to mitigate its impact on patients undergoing chemotherapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of non-metastatic breast cancer
* Indication for neoadjuvant or adjuvant chemotherapy as part of standard clinical practice
* Chemotherapy-naïve patients (no chemotherapy received in the previous 12 months)
* Signed written informed consent

Exclusion Criteria:

* Terminal or metastatic disease
* Pre-existing taste or smell disorders (e.g., anosmia, dysgeusia, neurological syndromes, etc.)
* Known allergies to any substances used in taste and chemesthetic function tests (e.g., quinine dihydrochloride, monosodium L-glutamate, capsaicin, etc.)
* Receiving neoadjuvant or adjuvant chemotherapy within research protocols
* Lack of signed written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This group includes male and female participants diagnosed with non-metastatic breast cancer who are receiving neoadjuvant or adjuvant chemotherapy according to standard clinical practice. Participants are treated at the Oncology Unit of Michele and Pietro Ferrero Hospital in Verduno. Eligible participants are those for whom chemotherapy is indicated as part of their routine care, and who are willing and able to complete sensory tests, nutritional assessments, and quality of life questionnaires during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dysgeusia during chemotherapy | - Baseline: within 15 days before the start of chemotherapy - Mid-treatment: approximately 3 months after baseline - End of chemotherapy: within 15 days after the completion of chemotherapy - Follow-up: 2 months after the end of chemotherapy
  The primary endpoint is the incidence of dysgeusia after the start of chemotherapy in participants with non-metastatic breast cancer. Taste perception will be evaluated using standardized taste strips to determine recognition thresholds for four basic tastes (sweet, sour, salty, and bitter). Dysgeusia will be considered present if the total taste strip score is lower than 9 at any of the evaluated time points.

SECONDARY OUTCOMES:
Quantitative changes in taste recognition thresholds | - Baseline: within 15 days before the start of chemotherapy - Mid-treatment: approximately 3 months after baseline - End of chemotherapy: within 15 days after completion of chemotherapy - Follow-up: 2 months after the end of chemotherapy
  Quantitative evaluation of recognition thresholds for the five basic tastes (sweet, sour, salty, bitter, and umami) to assess changes in taste perception during and after chemotherapy.
Chemesthetic sensitivity assessed by capsaicin strips | - Baseline: within 15 days before the start of chemotherapy - Mid-treatment: approximately 3 months after baseline - End of chemotherapy: within 15 days after completion of chemotherapy - Follow-up: 2 months after the end of chemotherapy
  Evaluation of chemesthetic function using strips impregnated with capsaicin at four increasing concentrations to assess oral sensitivity to chemical stimuli.
Taster status assessment | - Baseline: within 15 days before the start of chemotherapy - Mid-treatment: approximately 3 months after baseline - End of chemotherapy: within 15 days after completion of chemotherapy - Follow-up: 2 months after the end of chemotherapy
  Assessment of participants' "taster status" (ability to detect bitter compounds) to evaluate its potential correlation with the subsequent development of dysgeusia.
Chemotherapy-induced taste alteration (CiTAS) questionnaire | - Baseline: within 15 days before the start of chemotherapy - Mid-treatment: approximately 3 months after baseline - End of chemotherapy: within 15 days after completion of chemotherapy - Follow-up: 2 months after the end of chemotherapy
  Evaluation of participant-reported taste alterations using the Chemotherapy-Induced Taste Alteration Scale (CiTAS) and comparison with objective sensory test findings.
  Score range: 1 to 5. Higher scores indicate more severe taste alterations.
Nutritional status assessment | - Baseline: within 15 days before the start of chemotherapy - Mid-treatment: approximately 3 months after baseline - End of chemotherapy: within 15 days after completion of chemotherapy - Follow-up: 2 months after the end of chemotherapy
  Evaluation of nutritional status using the Global Leadership Initiative on Malnutrition (GLIM) criteria and measurement of phase angle using bioelectrical impedance analysis (BIA).
Caloric and macronutrient intake | - Baseline: within 15 days before the start of chemotherapy - Mid-treatment: approximately 3 months after baseline - End of chemotherapy: within 15 days after completion of chemotherapy - Follow-up: 2 months after the end of chemotherapy
  Assessment of caloric and macronutrient intake using 24-hour dietary recall interviews to determine changes during and after chemotherapy.
Quality of life assessment (FACT-G) | - Baseline: within 15 days before the start of chemotherapy - Mid-treatment: approximately 3 months after baseline - End of chemotherapy: within 15 days after completion of chemotherapy - Follow-up: 2 months after the end of chemotherapy
  Evaluation of quality of life using the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire.
  The total score is derived by summing scores from four domains (physical, social/family, emotional, and functional well-being). Each item is scored on a 5-point scale from 0 ("Not at all") to 4 ("Very much").

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sawicki CM, Janal MN, Nicholson SJ, Wu AK, Schmidt BL, Albertson DG. Oral cancer patients experience mechanical and chemical sensitivity at the site of the cancer. BMC Cancer. 2022 Nov 11;22(1):1165. doi: 10.1186/s12885-022-10282-3. PMID 36368973
- [Background] Turcott JG, Juarez-Hernandez E, De la Torre-Vallejo M, Sanchez-Lara K, Luvian-Morales J, Arrieta O. Value: Changes in the Detection and Recognition Thresholds of Three Basic Tastes in Lung Cancer Patients Receiving Cisplatin and Paclitaxel and Its Association with Nutritional and Quality of Life Parameters. Nutr Cancer. 2016;68(2):241-9. doi: 10.1080/01635581.2016.1144075. Epub 2016 Mar 4. PMID 26943275
- [Background] Epstein JB, de Andrade E Silva SM, Epstein GL, Leal JHS, Barasch A, Smutzer G. Taste disorders following cancer treatment: report of a case series. Support Care Cancer. 2019 Dec;27(12):4587-4595. doi: 10.1007/s00520-019-04758-5. Epub 2019 Mar 29. PMID 30927113
- [Background] Nolden AA, Hwang LD, Boltong A, Reed DR. Chemosensory Changes from Cancer Treatment and Their Effects on Patients' Food Behavior: A Scoping Review. Nutrients. 2019 Sep 24;11(10):2285. doi: 10.3390/nu11102285. PMID 31554217
- [Background] Landis BN, Welge-Luessen A, Bramerson A, Bende M, Mueller CA, Nordin S, Hummel T. "Taste Strips" - a rapid, lateralized, gustatory bedside identification test based on impregnated filter papers. J Neurol. 2009 Feb;256(2):242-8. doi: 10.1007/s00415-009-0088-y. Epub 2009 Feb 7. PMID 19221845
- [Background] Mueller CA, Pintscher K, Renner B. Clinical test of gustatory function including umami taste. Ann Otol Rhinol Laryngol. 2011 Jun;120(6):358-62. doi: 10.1177/000348941112000602. PMID 21774441
- [Background] Mueller C, Kallert S, Renner B, Stiassny K, Temmel AF, Hummel T, Kobal G. Quantitative assessment of gustatory function in a clinical context using impregnated "taste strips". Rhinology. 2003 Mar;41(1):2-6. PMID 12677732
- [Background] Buttiron Webber T, Briata IM, DeCensi A, Cevasco I, Paleari L. Taste and Smell Disorders in Cancer Treatment: Results from an Integrative Rapid Systematic Review. Int J Mol Sci. 2023 Jan 28;24(3):2538. doi: 10.3390/ijms24032538. PMID 36768861